CLINICAL TRIAL: NCT04808336
Title: Platelet Rich Plasma Injection Versus Surgical Fixation Procedure in Management of Spondylolisthesis grade1.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Dalia Salah Saif, lecturer of Rheumatology at faculty of medicine Menoufia University, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19719NEUS6
Record Dates: First submitted 2021-03-14; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Degenerative Spondylolisthesis G1

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP injection group (Active Comparator): Group 1: thirty patients were injected in the facet joint capsule with a series of three ultrasound-guided PRP injections at four-week intervals,
  Interventions: Other: PRP injection.
- surgical group.. (Active Comparator): Group 2: thirty patients underwent surgery
  Interventions: Procedure: fixation surgical procedure

INTERVENTIONS:
Other: PRP injection. — Group 1: thirty patients were injected in the facet joint capsule with a series of three ultrasound-guided PRP injections at four-week intervals,
  Arms: PRP injection group
Procedure: fixation surgical procedure — Group 2: thirty patients underwent surgery
  Arms: surgical group..

SUMMARY:
Spondylolisthesis is a serious health condition that is often treated with surgery or pain-relieving lumbar epidural steroids. Patients with persistent and debilitating symptoms who have failed to respond to conservative treatment should consider surgery.

Objectives: The aim of this study was to compare the therapeutic efficacy of three ultrasound guided PRP injections of the facet joint capsule to surgical procedures in patients with degenerative spondylolisthesis G1 and their effect on neurogenic pain relief and functional improvement over a one-year follow-up period.

Methods:

A one-year prospective randomised comparative clinical trial was performed on 60 patients with degenerative spondylolisthesis G1 who were randomly assigned to one of two groups: Group 1: thirty patients were injected in the facet joint capsule with a series of three ultrasound-guided PRP injections at four-week intervals, and Group 2: thirty patients underwent surgery. They were exposed to clinical neuropsychological testing.They were assessed for pain and function using clinical neurological assessments, VAS (Visual Analogue Scale), FRI (Functional Rating Index), Roland Morris, and ODI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with degenerative spondylolithesis Grade 1 were diagnosed based on their clinical and radiological image.
* Patients complained of extreme pain and received medical treatment (NSAIDS) without improvement.

Exclusion Criteria:

* Patients with more than two-level pathological lesions and those who had previously
* Patients undergone lumbar surgery,
* HCV, HBV infected patients,
* patients with local abscesses,
* diabetes mellitus,
* malignancy, pregnancy,
* blood disorders (coagulopathy, thrombocytopenia),
* patients who had previously received local injection of steroid within past 3 weeks
* Patients who had undergone lumbar surgery,
* patients with advanced spondylolithesis, disc prolapse,
* inflammatory or musculoskeletal disorders of the spine.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2020-05-02 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
1-Visual analogue scale. , | 12 months
  VAS Visual analogue scale: According to the VAS, the pain severity was calculated by the patients on a scale of 0 (no pain) to 10 (agonising pain)
2-The Persian Functional Rating Index (FRI ) | 12 months
  The Persian Functional Rating Index (FRI ), which is an accurate and valid instrument that contains 10 items that measure both pain and function, with an impairment score ranging from 0% (no disability) to 100% (severe disability) 2- The Persian Functional Rating Index (FRI ), which is an accurate and valid instrument that contains 10 items that measure both pain and function, with an impairment score ranging from 0% (no disability) to 100% (severe disability)

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) for low back pain | 12 months
  Assessment of pain-related disability using the Oswestry Disability Index (ODI) for low back pain, which categorises disability as minimal (0-20), mild (20-40), extreme (40-60), ODI of 60-80 suggests that the patient is crippled, and ODI of 80-100 implies that the patient is either bed-ridden or exaggerating his or her complaints
The Roland-Morris questionnaire | 12 months
  The Roland-Morris questionnaire is a 24-item self-report checklist that assesses the extent at which low-back pain affects daily activities. Since each question is implies one point, scores will range from 0 (no disability) to 24 (severe disability)

CONTACTS AND LOCATIONS:
Locations (1):
- Dalia Saif, Shebien Elkom, Egypt